CLINICAL TRIAL: NCT03120572
Title: Effect of Concurrent Chemoradiation Therapy on Respiratory Muscle Performance, Lung Function and Functional Capacity in Patients With Local Esophagus Cancer
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Jen Chen, VS. Division of Radiation Oncology, Department of Radiology, Mackay Memorial Hospital
Other Study IDs: 11MMHIS183
Record Dates: First submitted 2017-03-14; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Esophageal Cancer
Keywords: Respiratory muscle strength; Diaphragmatic surface electromyography; Functional capacity
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months

SUMMARY:
The purpose of this study is to investigate the effect of concurrent chemoradiation therapy on respiratory muscle performance, lung function and functional capacity in patients with local esophagus cancer.

DETAILED DESCRIPTION:
This is a prospective observational study design. A total of 45 patients with newly diagnosed esophageal cancer will be recruited from the Mackay Memorial Hospital. All tests will be performed at baseline (prior to cancer treatment), weekly during treatment, prior to surgery, and one month after surgery. Tests will include demographic data collection, respiratory muscle performance (maximal inspiratory and expiratory pressure tests combined with diaphragmatic surface electromyography, and pulmonary functional test), dyspnea, and the functional exercise test (6-min walk test).Repeated measure ANOVA will be used for analyzing difference of parameters among various time points.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed primary esophageal cancer, aged more than 20 years, and communicate without difficulty

Exclusion Criteria:

* inability to perform inspiratory muscle training, the presence of unstable angina or myocardial infarction in recently one month, cannot cooperate with training protocols, and pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed primary esophageal cancer
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change of maximal inspiratory pressure (MIP) | Baseline, weekly during treatment, and 2 weeks after the completion of treatment
  Change from baseline MIP at the end of each week's treatment, and 2 weeks after the completion of treatment
Change of diaphragmatic surface electromyography (EMGdi) | Baseline, weekly during treatment, and 2 weeks after the completion of treatment
  Change from baseline EMGdi at the end of each week's treatment, and 2 weeks after the completion of treatment
Change of forced expiratory volume in one second (FEV1) | Baseline, weekly during treatment, and 2 weeks after the completion of treatment
  Change from baseline FEV1 at the end of each week's treatment, and 2 weeks after the completion of treatment
Change of forced vital capacity (FVC) | Baseline, weekly during treatment, and 2 weeks after the completion of treatment
  Change from baseline FVC at the end of each week's treatment, and 2 weeks after the completion of treatment

SECONDARY OUTCOMES:
Change of functional exercise capacity | Baseline, weekly during treatment, and 2 weeks after the completion of treatment
  Change from baseline 6-minute walking distance at the end of each week's treatment, and 2 weeks after the completion of treatment
Change of dyspnea | Baseline, weekly during treatment, and 2 weeks after the completion of treatment
  Change from baseline Modified Borg Dyspnea score at the end of each week's treatment, and 2 weeks after the completion of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan